CLINICAL TRIAL: NCT04139681
Title: Open Clinical Trial to Assess Safety and Efficacy of the Sore Throat Lozenges in Patients With Acute Sore Throats
Brief Title: Safety and Efficacy of the Sore Throat Lozenges to Treat Acute Sore Throats
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5'000'196
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Tonsillopharyngitis; Respiratory Tract Infection Viral

STUDY DESIGN:
Intervention Model Description: Eligible patients fulfilling the inclusion criteria will :
  1. First suck under supervision in the study centre one lozenge and document every 15 minutes the pain on a 100mmVAS for 90 minutes
  2. Receive the rest of the bottle still containing 19 lozenges and have to take them for 4 days (5 lozenges per day). The patients have to fill out a diary in the morning and in the evening filling out the Tonsillopharyngitis Score (TSS), pain on a 100mm VAS and occurrence of adverse events, intake of other medication.
  3. After the end of the treatment period patients will return to the study centre for the final visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A. Vogels Sore Throat Lozenges (Experimental): Each patients receives 1 glass containing 20 A.Vogel Sore Throat lozenges at inclusion visit 1. They first suck under supervision in the study centre one Vogel Sore Throat lozenge and document every 15 minutes the pain 90 minutes. Patients will receive the rest of the bottle still containing 19 Vogel Sore Throat lozenges and have to take them for 4 days (5 lozenges per day, throughout the day) and record tonsillitis pain.
  Interventions: Drug: A. Vogels Sore Throat lozenges

INTERVENTIONS:
Drug: A. Vogels Sore Throat lozenges — 5 times 1 A. Vogels sore throat lozenges daily for 4 days
  Other Names: Sore Throat lozenges

SUMMARY:
Aim of this study is to investigate safety and efficacy of A. Vogel Sore throat lozenges for the treatment of of acute sore throats

DETAILED DESCRIPTION:
75 patients aged 12-75 years with acute sore throats (symptoms not older than 48 h) were recruited by the study site/CRO via local general practitioners and are allocated to acute treatment with A. Vogel Sore throat lozenges. The patients who are confirmed to meet the study entry criteria and after having given written informed consent will be assigned to receive a study treatment according to study procedures described in the study plan.

The patients will visit study site twice. At the first visit (Visit 1) a screening will be performed to finally decide if patient will be included/excluded in the study. Then he or she will be taking one single lozenge under supervision of the investigating physician and acute efficacy/safety ratings recorded before intake and repeatedly every 15 minutes for 90 minutes after intake of first lozenge. He or she will be supplied with the remaining 19 lozenges in a bottle and provided with patient diaries for home recording of efficacy/safety. After four days (max 5 days) or until complete resolution of symptoms the patients were obliged to return to the study centre for final visit 2. Daily ratings of efficacy/safety was done by the patient once in the morning and once in the evening. Daily dosage was 5 lozenges per day every 3rd hour during daytime.

At final visit 2, patients will be evaluated physically by the physician at the study centre and again assessed for safety/efficacy parameters. At last, patients returned their patient diaries and remaining study medication before compensation is handed out and patients finally excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 12-75 years
* Acute pharyngitis or tonsillitis with the following symptoms: Sore throat, Inflammation of the pharynx and/or tonsils
* Start of painful disease with the last 48 hours before study inclusion
* Tonsillopharyngitis Score bigger than or equal to 6 (s.attachment)
* Willingness to give blood samples and three viral throat swabs
* Written informed consent

Exclusion Criteria:

* Pharyngitis or tonsillitis more than 48 hours before study start (inclusion)
* Intake of analgetically active medication within the last 12 hours prior to study start (inclusion)
* Use of local sore throat medications within the last 4 hours prior to study start (inclusion)
* Patients with symptoms of a primary bacterial pharyngitis or a bacterial superinfection
* Severe medical condition (tumors, uncontrolled hypertension, heart insufficiency, immunosuppressive diseases etc.)
* Systemic use of corticosteroids in the last month prior to study inclusion
* Allergies to substances used in the tablet
* Pregnancy or lactation
* Participation or inclusion in one or more clinical trials within the last 30 days

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Rate of "good" and "very good" tolerability ratings vs. "moderate" and "bad" tolerability ratings as assessment by a physician | 4 days
  Assessment of safety after acute intake of 90 minutes at visit 1 and after 4 days of continous intake at final visit 2 by physician with very good, good, moderate, bad

SECONDARY OUTCOMES:
Change of acute throat pain on a visual analog scale (VAS) | 90 min
  Change of acute throat pain (pain reduction) on a visual analog scale (VAS) ranging from 0 millimeters (no pain) to 100 millimeters (most severe pain) within 90 minutes compared to baseline
Rate and number of treatment responders at day 1,2,3,4 | 4 days
  Rate and number of Treatment responders expressed on a Tonsillopharyngitis Score (TSS) measuring change of sore throat symptoms at day 1,2,3,4 (Responder=TSS reduction by 50% compared to baseline). The TSS score consists the following four symptoms: throat pain, difficulty in swallowing, salivation, reddening and fever (fever was defined as >38.5°C for this score) which are all rated on a scale with 0=none, 1=mild, 2=moderate, 3=severe.
Total change of Tonsillopharyngitis Score (TSS) at the end of treatment | 4 days
  Change of Tonsillopharyngitis Score (TSS) total at the end of treatment at day 4 as compared to baseline measurement. The TSS score consists the following four symptoms: throat pain, difficulty in swallowing, salivation, reddening and fever (fever was defined as >38.5°C for this score) which are all rated on a scale with 0=none, 1=mild, 2=moderate, 3=severe.
Total reduction of pain score | 4 days
  Change of acute throat pain (pain reduction) on a visual analog scale (VAS) ranging from 0 millimeters (no pain) to 100 millimeters (most severe pain) on the evenings of day 1,2,3,4 compared to baseline
Absolute and relative distribution of individual Tonsillopharyngitis Score (TSS) symptoms | 4 days
  Absolute and relative distribution of the single symptoms: throat pain, difficulty in swallowing, salivation, reddening and fever (fever was defined as >38.5°C for this score) from the Tonsillopharyngitis Score (TSS) on day 1,2,3,4 compared to baseline
The relative number of painfree patients | 4 days
  The relative number of painfree patients that experience a change of acute throat pain (pain reduction) on a visual analog scale (VAS) ranging from 0 millimeters (no pain) to 100 millimeters (most severe pain) of lower than 10 (<10) at day 1,2,3,4 compared to baseline
The average time taken to symptom resolution1 | 4 days
  The time taken to symptom resolution reaching a Tonsillopharyngitis Score (TSS) of less than 3 (<3). The TSS score consists the following four symptoms: throat pain, difficulty in swallowing, salivation, reddening and fever (fever was defined as >38.5°C for this score) which are all rated on a scale with 0=none, 1=mild, 2=moderate, 3=severe.
The average time to symptom resolution2 | 4 days
  The average time required for subjective symptom resolution
The rate and kind of concomitant medication use | 4 days
  The rate of use and kind of concomitant medication that are used by patients are recorded by questionaire as part of the patient diary and analyzed in descriptive manner
The throat status as assessed by the investigating physician | 4 days
  Throat status (reddening, swelling, inflammation) assessed by physician. Assessed are: The presence of reddening in the throat (yes/no) and swelling (light, moderate, severe) and reddening, swelling, and coating of the tonsils (yes/no). beginning vs. after 90 minutes of treatment vs. 4 days of treatment.
Rate of "good" and "very good" efficacy ratings vs. "moderate" and "bad" efficacy ratings as assessment by a 1) physician 2) the patient | 4 days
  Global subjective assessment of the subjective efficacy after acute intake of 90 minutes at visit 1 and after 4 days of continous intake at final visit 2 rated 1) by physician and 2) by the patient with "very good", "good", "moderate", "bad"
Rate of treatment acceptance (yes) by the patient | 4 days
  The rate of treatment acceptance assessed by asking patients if they would retake the IMP (yes) or refuse (no) at final visit 2.
The rate and kind of occuring adverse events | 4 days
  The rate and kind of occuring adverse events assessed at visit 2 and analyzed in descriptive manner
Rate of "good" and "very good" tolerability ratings vs. "moderate" and "bad" efficacy ratings as assessment by the patient | 4 days
  Global subjective assessment of the subjective tolerability after acute intake of 90 minutes at visit 1 and after 4 days of continous intake at final visit 2 rated by the patient with "very good", "good", "moderate", "bad"
Rate and kind of clinically relevant changes in vital parameters as assed by physical examination by the investigating physician | 4 days
  Rate and kind of clinically relevant changes in vital parameters (pulse, both blood pressure, body temperature) derived from exhamination by investigating physician at inclusion visit 1 and at final visit 2
Rate and kind of clinically relevant changes in blood parameters examined by the investigating physician | 4 days
  Rate and kind of clinically relevant changes in blood parameters measured from haematological and biochemical analysis of blood samples analyses as asssessed by the investigating physician. Laboratory blood values that are measured: ALAT, ASAT, total bilirubin, plasma glucose, serum creatinine, ESR (1h), CRP, total cholesterol, erythrocytes, MCHC, MCH, MCV, hematocrit, hemoglobin, leukocytes, and thrombocytes] derived from clinical laboratory analyses and assessed by investigating physician at visit 1 and compared to measurements at final visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Alexandar Buchkov, Dr. med., Principal Investigator — Diagnostics and Consultation Center Convex
Locations (1):
- Diagnostics and Consultation Center Convex EOOD, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No